CLINICAL TRIAL: NCT03593915
Title: A Phase 1b/2, Open-label Clinical Study to Determine Preliminary Safety and Efficacy of Alvocidib When Administered in Sequence After Decitabine or Azacitidine in Patients With MDS
Brief Title: A Phase 1b/2 Study of Alvocidib Plus Decitabine or Azacitidine in Patients With MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor decided not to continue the study based on the overall company strategy in AML.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI-ALV-102
Record Dates: First submitted 2018-05-24; First posted 2018-07-20 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Previously untreated MDS; MDS who have received <6 cycles of treatment with hypomethylating agents (HMAs); De novo or secondary MDS (treatment-related) who are not eligible for intensive induction chemotherapy or stem cell transplant; FAB subtypes: refractory anemia [RA], RA w/ ringed sideroblasts, RA w/ excess blasts, RA w/ excess blasts in transformation or chronic myelomonocytic leukemia; Intermediate and above per the Revised International Prognostic Scoring System (IPSS-R) groups; Sumitomo Oncology SMPO; Cancer; Phase 1b/2
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Neoplasms | interventions — alvocidib; Decitabine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ph 1b and 2: MDS (Experimental): * Patients with previously untreated MDS
  * Patients with MDS who have received <6 cycles of HMAs (during dose escalation only)
  * Patients with de novo (cause unknown) or secondary MDS (treatment-related) who are not eligible for intensive induction chemotherapy or stem cell transplant
    * All French-American-British (FAB) subtypes
    * Intermediate and above per IPSS-R groups
  Interventions: Combination Product: Alvocidib Plus Decitabine (during dose escalation only) or Azacitidine

INTERVENTIONS:
Combination Product: Alvocidib Plus Decitabine (during dose escalation only) or Azacitidine — PHASE 1b:
  Decitabine administered as an intravenous (IV) infusion daily for 5 days at a dose of 20 mg/m2 followed on Day 8 by alvocidib as a loading dose over 30 minutes followed by a 4-hour IV infusion (hybrid dosing) Once the maximum dose of alvocidib administered via hybrid dosing has been determined, 2 cohorts of patients will receive azacitidine followed by alvocidib administered as an IV infusion. Azacitidine may be administered as either an IV bolus over 10 to 40 minutes or as a subcutaneous (SC) injection on either a 7 day or 5-2 2 schedule. Regardless of which azacitidine schedule or route of administration is used, alvocidib will be given on Day 10 as a 30-to-60 minute IVI
  PHASE 2:
  The Phase 2 study will use the RP2D from the Phase 1b study and follow a Simon 2-stage minimax design using the RP2D of alvocidib administered as a 30-to-60 minute IV infusion determined in the Ph1b study to explore efficacy of alvocidib when administered in sequence after azacitidine.

SUMMARY:
Alvocidib, a cyclin-dependent kinase 9 (CDK 9) inhibitor, in time-sequential therapy demonstrated significant clinical activity in secondary AML patients with prior MDS. Patients with IPSS-R intermediate and above MDS have an increased risk of developing AML and may be treated with the same chemotherapy regimens used in patients with AML. Eight Phase I or II clinical trials have been completed in patients with AML, totaling more than 400 patients with both relapsed/refractory or newly diagnosed AML.

Preclinical studies have demonstrated that decitabine exposure increased the expression of NOXA, which is a specific antagonist of the survival factor MCL 1. Pharmacologic downregulation of MCL-1 via CDK 9 inhibition, as well as upregulation of the MCL-1 antagonist, NOXA, following decitabine exposure may result in enhanced antileukemic activity in MCL-1-dependent malignancies.

DETAILED DESCRIPTION:
PHASE 1b:

Patients will be enrolled in cohorts of 3-6 patients. Escalation of the alvocidib dose will follow a standard 3+3 design with sequential cohorts of 3 patients treated with incrementally higher doses of alvocidib administered in sequence after decitabine (during dose escalation) or azacitidine until a dose-limiting toxicity (DLT) is observed and the MTD is established.

Once the MTD or preliminary RP2D of alvocidib administered via hybrid dosing is identified, 2 cohorts of at least 3 patients each will receive azacitadine followed by alvocidib administered as a 30-60 minute IV infusion.

Expansion at MTD Once the MTD or preliminary RP2D of alvocidib administered as a 30-to-60 minute IV infusion is determined, up to 25 patients will be enrolled in an Expansion cohort to receive alvocidib following azacitadine to confirm safety, explore potential biomarkers, and evaluate potential signals of alvocidib activity. Once this Expansion cohort is completed, the study will progress to Phase 2

PHASE 2:

Phase 2 design is based on the Simon 2-stage minimax design (Simon 1989).

* Stage 1: Up to 15 evaluable patients will be enrolled and treated at the RP2D identified in the Phase 1b study.
* Stage 2: Ten patients will be enrolled to bring the total enrollment in Phase 2 (including Stage-1 patients) to 25 evaluable patients. Stage-2 patients will also receive the RP2D dose of alvocidib administered by 30-to-60 minute IV infusion identified in the Phase 1b study. If 6 or more responses are observed in 25 patients, the conclusion will be that the combination regimen is worthy of further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. Phase 1b Dose Escalation: Patients with previously untreated MDS and patients with MDS who received fewer than six (6) cycles of previous HMAs. Phase 1b Expansion: Untreated patients with de novo or secondary MDS. Phase 2: Untreated patients with de novo or secondary MDS
3. Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score ≤2 at enrollment
4. Provide written informed consent prior to any study-related procedure. (In the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed.)
5. Patients with a life expectancy of ≥3 months (90 days)
6. Patients with adequate major organ functions meeting the following criteria on the basis of laboratory data within 4 weeks (28 days) before enrollment (if multiple data are available, most recent data during the period):

   1. Serum creatinine: ≤1.8× the upper limit of the normal (ULN) range
   2. Total bilirubin: ≤2× the ULN
   3. Aspartate transaminase (AST) and alanine transaminase (ALT): ≤3× the ULN
   4. Left ventricular ejection fraction (LVEF) >45% by echocardiogram or multigated acquisition (MUGA) scan
7. Be able to comply with the requirements of the entire study.
8. Patients with Revised International Prognostic Scoring System (IPSS-R) intermediate-, high-, and very high-risk MDS

Exclusion Criteria:

1. Presence of concomitant severe cardiovascular disease:

   1. Patients who had myocardial infarction within 6 months (180 days) before enrollment
   2. Patients with significant diseases at enrollment that may affect study treatment, such as New York Heart Association (NYHA) Functional Class III or IV heart disease, National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade ≥3 arrhythmia, angina pectoris, abnormal electrocardiogram findings, interstitial pneumonia or pulmonary fibrosis
2. Presence of concomitant malignancy requiring chemotherapy or any malignancy (except basal and squamous cell carcinoma of the skin) for which the patient received chemotherapy within 6 months prior to enrollment. NOTE: Diagnosis of any previous or concomitant malignancy is thus not an exclusion criterion.
3. Presence of uncontrolled or uncontrollable infection(s); or ≥Grade 3 infection according to NCI CTCAE v5.0
4. Presence of any psychological, familial, sociological or geographical condition that, in the opinion of the investigator, could potentially hinder compliance with the study protocol and follow-up schedule
5. Patients with a dry tap on bone marrow aspiration before enrollment
6. Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease, or patients who require long-term systemic steroid therapy greater than the equivalent of 20 mg of prednisone daily (excluding therapy given on an 'as needed' [PRN] basis)
7. Patients with other documented malignancies within past year aside from synchronous or metachronous multiple cancers with a disease-free period of ≤5 years (excluding carcinoma in situ, mucosal carcinoma, or other such carcinomas curatively treated with local therapy)
8. Patients with ≥Grade 2 hemorrhage according to NCI CTCAE v5.0
9. Patients who have previously received alvocidib or another cyclin-dependent kinase 9 (CDK9) inhibitor
10. Patients who are pregnant or breastfeeding
11. Female patients of childbearing potential who are sexually active and unwilling to use a medically acceptable method of contraception associated with a low failure rate prior to study entry, for the duration of study participation and for at least 6 months after the last dose of study drug. (Patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy, or bilateral tubal ligation / salphingectomy, or postmenopausal for at least 2 years.)
12. Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second effective method of contraception during the trial and for at least 3 months after the last administration of study treatment.
13. Patients who are inappropriate for participation in the study for other reasons in the opinion of the investigator or sub-investigator(s)
14. Patients with a known hypersensitivity to decitabine (those patients enrolled in escalation) or azacitidine or mannitol
15. Patients who have received erythropoietin-stimulating agents (ESAs) within 2 weeks (14 days) prior to Cycle 1/Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anthony, DO, Study Director — Sumitomo Pharma America, Inc.
Locations (12):
- United States (12):
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - US Oncology - Texas Oncology - Austin Midtown, Austin, Texas
  - US Oncology - Texas Oncology - Baylor University Medical Center, Dallas, Texas
  - US Oncology - Texas Oncology - Fort Worth, Fort Worth, Texas
  - US Oncology - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - US Oncology - Texas Oncology - Tyler, Tyler, Texas
  - US Oncology - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - US Oncology - Northwest Cancer Specialists, P.C., Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty subjects were enrolled between August 2018 and August 2021
Pre-assignment Details: In phase 1b, patients were enrolled in cohorts of 3-6 patients. Escalation of alvocidib (ALV) dose followed standard 3+3 dosing with sequential cohorts of 3 patients treated at incrementally higher doses of alvocidib administered in sequence after fixed doses of decitabine (DEC) or azacitadine (AZA) until MTD is reached.
Groups:
- ALV-DEC: Cohort 1: Decitabine is administered as a 1-hour intravenous (IV) infusion (IVI) daily days 1-5 at 20mg/m2; followed on day 8 by Alvocidib 20mg/m2 (30min bolus) and Alvocidib 20mg/m2 (4 hr IVI)
- ALV-DEC: Cohort 2: Decitabine is administered as a 1-hour intravenous (IV) infusion (IVI) daily days 1-5 at 20mg/m2; followed on day 8 by Alvocidib 20mg/m2 (30min bolus) and Alvocidib 30mg/m2 (4 hr IVI)
- ALV-DEC: Cohort 3: Decitabine is administered as a 1-hour intravenous (IV) infusion (IVI) daily days 1-5 at 20mg/m2; followed on day 8 by Alvocidib 20mg/m2 (30min bolus) and Alvocidib 45mg/m2 (4 hr IVI)
- ALV-DEC: Cohort 4: Decitabine is administered as a 1-hour intravenous (IV) infusion (IVI) daily days 1-5 at 20mg/m2; followed on day 8 by Alvocidib 20mg/m2 (30min bolus) and Alvocidib 60mg/m2 (4 hr IVI)
- ALV-AZA: Cohort 5: Azacitidine (AZA) administered on either a 7-day schedule or a 5-2-2 schedule (once daily for 5 days followed by 2 drug-free days with 2 more days of treatment) at 75mg/m2 per day subcutaneously or via IVI. Alvocidib (ALV) administered on day 10 at 75mg/m2 as a 30-60 minute IVI.
- ALV-AZA: Cohort 6: Azacitidine (AZA) administered on either a 7-day schedule or a 5-2-2 schedule (once daily for 5 days followed by 2 drug-free days with 2 more days of treatment) at 75mg/m2 per day subcutaneously or via IVI. Alvocidib (ALV) administered on day 10 at 90mg/m2 as a 30-60 minute IVI.
Period: Overall Study
Arm/Group | ALV-DEC: Cohort 1 | ALV-DEC: Cohort 2 | ALV-DEC: Cohort 3 | ALV-DEC: Cohort 4 | ALV-AZA: Cohort 5 | ALV-AZA: Cohort 6
Started (Any patient who received at least 1 dose of study drug.) | 3 | 3 | 3 | 4 | 3 | 4
Completed (Completed Cycle 1) | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALV-DEC: Cohort 1 | ALV-DEC: Cohort 2 | ALV-DEC: Cohort 3 | ALV-DEC: Cohort 4 | ALV-AZA: Cohort 5 | ALV-AZA: Cohort 6 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 4 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 0 | 2 | 0 | 0 | 4
  >=65 years | 3 | 1 | 3 | 2 | 3 | 4 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 0 | 2 | 9
  Male | 2 | 1 | 2 | 1 | 3 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 3 | 3 | 3 | 3 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Assessment of safety of alvocidib administered in combination with either decitabine (DEC) or azacitidine (AZA) by reporting of adverse events and serious adverse events
Time Frame: From the time of first dose to 30 days after the last dose, an average of 33.7 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | ALV-DEC: Cohort 1 | ALV-DEC: Cohort 2 | ALV-DEC: Cohort 3 | ALV-DEC: Cohort 4 | ALV-AZA: Cohort 5 | ALV-AZA: Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 4
Participants | 3 | 3 | 3 | 4 | 3 | 4

2. Primary Outcome: Tolerability of Alvocidib as Evaluated by Incidence of Dose Limiting Toxicities (DLTs) as Observed in Cycle 1
Description: The DLTs are defined as follows based on the NCI CTCAE v5.0: Must be at least possibly related to Alvocidib; Any Gr 4 nonhematologic toxicity; Gr 3 nonhematologic toxicity that does not resolve to ≤Gr 2 in 48 hours; Gr 3 diarrhea, mucositis, nausea, or vomiting will be considered dose limiting only if resolution to ≤Gr 2 requires >7 days; and ≥Grade 3 creatinine elevation that does not resolve to <G2 within 7 days.
Time Frame: Cycle 1 (28 days)
Population: Sponsor's decision to terminate further development of the alvocidib program. Data collection and analysis were therefore not conducted as planned.
Arm/Group | ALV-DEC: Cohort 1 | ALV-DEC: Cohort 2 | ALV-DEC: Cohort 3 | ALV-DEC: Cohort 4 | ALV-AZA: Cohort 5 | ALV-AZA: Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Determination of the Complete Response Rate
Description: The calculation for Complete Response Rate is as follows: complete response [CR] / complete response with incomplete blood count recovery [CRi] / CRmarrow / partial response [PR] / hematologic improvement [HI]
Time Frame: From the date of first treatment, every 8 weeks, for the first 6 cycles, for an average of 26 weeks
Population: as for outcome 2
Arm/Group | ALV-DEC: Cohort 1 | ALV-DEC: Cohort 2 | ALV-DEC: Cohort 3 | ALV-DEC: Cohort 4 | ALV-AZA: Cohort 5 | ALV-AZA: Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Improvement in Transfusion Dependence
Description: Determine if treatment with alvocidib administered in sequence after DEC or AZA resulted in improvements in transfusion dependence
Time Frame: Duration of study treatment up to 6 months
Population: Sponsor's decision to terminate further development of the alvocidib program. Data collection and analysis were not conducted as planned.
Arm/Group | ALV-DEC: Cohort 1 | ALV-DEC: Cohort 2 | ALV-DEC: Cohort 3 | ALV-DEC: Cohort 4 | ALV-AZA: Cohort 5 | ALV-AZA: Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, an average of 6 months.
Arm/Group | ALV-DEC: Cohort 1 | ALV-DEC: Cohort 2 | ALV-DEC: Cohort 3 | ALV-DEC: Cohort 4 | ALV-AZA: Cohort 5 | ALV-AZA: Cohort 6
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 4/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 1/3 | 3/4 | 3/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALV-DEC: Cohort 1 (N=3) | ALV-DEC: Cohort 2 (N=3) | ALV-DEC: Cohort 3 (N=3) | ALV-DEC: Cohort 4 (N=4) | ALV-AZA: Cohort 5 (N=3) | ALV-AZA: Cohort 6 (N=4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetes Insipidus (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALV-DEC: Cohort 1 (N=3) | ALV-DEC: Cohort 2 (N=3) | ALV-DEC: Cohort 3 (N=3) | ALV-DEC: Cohort 4 (N=4) | ALV-AZA: Cohort 5 (N=3) | ALV-AZA: Cohort 6 (N=4)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3 | 4 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 4 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 3 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Oral Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastri Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 2 | 2 | 3 | 1 | 3
Neutrophil Count Decreased (Investigations) | 1 | 1 | 1 | 2 | 2 | 2
White Blood Cell Count Decreased (Investigations) | 1 | 1 | 1 | 2 | 3 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 2 | 1 | 2 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 1 | 2 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 2 | 0 | 2 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Weight Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood Phosphorous Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Coronavirus Test Positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Serum Ferritin Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Troponin I Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 3 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 1 | 1 | 3
Non-cardiac Chest Pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Localised Oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Catheter Site Vesicles (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion Site Extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hypomagnasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 2 | 2 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Memory Impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Parasthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2 | 0
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Foreign Body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Vascular Access Complications (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Periorbial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1
Hot Flush (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scleral Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cancer Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Sinus Operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetes Insipidus (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Humerous Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
A business decision was made to stop enrollment and the study was discontinued on 17 November 2020. Consistent with Food and Drug Administration and International Council for Harmonisation guidance on the content for abbreviated and synoptic CSRs, only safety data are analyzed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT03593915/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT03593915/SAP_001.pdf